CLINICAL TRIAL: NCT06601582
Title: Effectiveness of a Intraoperative Blood Recovery System in Cardiovascular Surgery Using Cardiopulmonary Bypass in Brazil. Randomized Crontrolled Trial
Brief Title: Effectiveness of a Intraoperative Blood Recovery System in Cardiovascular Surgery in Brazil
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Livia Barboza de Andrade, Director of Education, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IMIFernandoFigueira
Record Dates: First submitted 2023-04-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Surgery; Blood Loss, Surgical
Keywords: Cardiovascular Surgery; Operative Blood Salvage
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Device: Use of a operative blood salvage system The surgical team will use a operative blood salvage system
  Interventions: Device: Use of a operative blood salvage system
- No intervention (No Intervention)

INTERVENTIONS:
Device: Use of a operative blood salvage system — The surgical team will use a operative blood salvage system
  Arms: Intervention

SUMMARY:
Randomized trial to evaluate the effectiveness of a intra operative blood recovery system in reducing the need for allogeneic transfusion in cardiovascular surgeries using cardiopulmonary bypass

DETAILED DESCRIPTION:
To evaluate the effectiveness of a intra operative blood recovery system in reducing the need for allogeneic transfusion in cardiovascular surgeries using cardiopulmonary bypass, a randomized clinical trial will be conducted. The study will be conducted at a teaching hospital, which is a reference for major cardiac surgeries and receives patients from the Brazilian Unified Health System (SUS). The patients will be randomly assigned to two groups: with and without the use of the system, and allocation concealment will be performed. Continuous variables will be analyzed through frequency distributions and appropriate descriptive measures (mean or median), while categorical variables will be presented through frequency distributions. For categorical variables, the confidence interval will be calculated, conventionally set at 95%. For continuous variables, the T-test will be used to measure differences, while for categorical variables, the McNemar statistical test will be used. For all analyses, a significance level of 5% will be used, and the data will be analyzed according to the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing CABG or Valve surgery singly.

Exclusion Criteria:

* Emergency cardiac surgery;
* Previous heart surgery;
* End-stage chronic kidney disease;
* Inability to receive a blood transfusion (refusal);
* Anemia (hemoglobin less than 10g/dl);
* Thrombocytopenia (platelet count less than 100,000/mm3);
* Coagulopathy (RNI > 1.5);

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years old and older
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood transfusion rate | 2 days
  Reduction in the volume of packed red blood cells administered intrao peratively

SECONDARY OUTCOMES:
Hospital mortality | 30 days
  Rate of Hospital mortality within 30 days
Hospital Stay | 30 days
  Number of Hospital stay in days
ICU stay | 30 days
  Number of ICU stay in days
Mechanical ventilation | 30 days
  Time of mechanical ventilation
Re-operation for bleeding | 30 days
  Rate of Re-operation for bleeding
Need for renal replacement therapy | 30 days
  Rate of Need for renal replacement therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Integral Medicine Institute Professor. Fernando Figueira-IMIP, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No